CLINICAL TRIAL: NCT06405763
Title: Snodgrass Versus Grafted Snodgrass Repair in Narrow Urethral Plate in Distal Penile Hypospadias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Shawky Gebaly, Resident doctor at urology department, Sohag university hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-12-06MS
Record Dates: First submitted 2024-04-28; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snodgrass repair group (Active Comparator): A relaxing incision is made in the midline by using scalpel or scissors from Within the meatus to the end of the plate.
  A 6 F stent is passed into the bladder. The neourethra is closed using a fine suture, 7-0 or 6-0 vicryl sutures in two-layer.
  Interventions: Procedure: Snodgrass repair
- Snodgrass repair with graft group (Active Comparator): A relaxing incision is made in the midline by using scalpel or scissors A free graft was measured and harvested from the inner prepuce and was defatted and sutured onto the incised urethral plate after the urethral plate was incised he graft was sutured overlying the incision line A 6 F stent is passed into the bladder. The neourethra is closed
  Interventions: Procedure: Snodgrass repair with graft

INTERVENTIONS:
Procedure: Snodgrass repair — A relaxing incision is made in the midline by using scalpel or scissors
  A 6 F stent is passed into the bladder. The neourethra is closed
  Arms: Snodgrass repair group
Procedure: Snodgrass repair with graft — A relaxing incision is made in the midline by using scalpel or scissors In grafted Snodgrass repairA free graft was measured and harvested from the inner prepuce and was defatted and sutured onto the incised urethral plate The graft was sutured overlying the incision line A 6 F stent is passed into the bladder. The neourethra is closed
  Arms: Snodgrass repair with graft group

SUMMARY:
We aime to compare between Snodgrass and grafted Snodgrass repair in the outcome in distal penile hypospadias with urethral plate less than 8mm

DETAILED DESCRIPTION:
The main goal for hypospadias repair is to achieve both cosmetic and functional normality.

Several surgical techniques for hypospadias repair have been developed that depend on the site of the urethral meatus in children The effect of the urethral plate characteristics on the surgical outcome of Snodgrass repair has been studied in many series. Some documented that urethral plate width has a significant impact on the complication rates Holland and Smith reported a high complication rate in Snodgrass repair with a urethral plate width of less than 8 mm 7 The augmentation of the urethral plate either with inlay graft (DIGU, Snodgraft, or G-TIP), Onlay preputial flap, or other flaps carries a better outcome than the original TIP in many studies Others denied any effect of the narrow urethral plate on the success rate We aim in this study to determine which is better in narrow urethral plate in distal penile hypospadias, as regarding surgical and cosmetic outcomes; Snodgrass or combined inner preputial graft with Snodgrass

ELIGIBILITY:
Inclusion Criteria:

Children age: > 6m up to 16y

* Distal penile hypospadias(distal shaft,coronal,subcoronal )
* mid penile hypospadias with mild chordae les 30 degree
* Urethral plate <8 mm in maximum transverse diameter before the midline urethral plate incision .Primary non-circumcised cases of hypospadias

Exclusion Criteria:

* Proximal and mid penile hypospadias with marked chordae
* previous hypospadias repair

Ages: 6 Months to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 12 months
  Investigators want to compare between Snodgrass and combined inner preputial graft with Snodgrass in functional outcome by evaluation of the stream an ideal stream of urine (single, compact, rifled, non-dispersed urinary stream of adequate caliber) without straining.
Cosmetic outcome | 12 months
  Investigators want to compare between Snodgrass and combined inner preputial graft with Snodgrass in cosmetic outcome By Hypospadias Objective penile Evaluation (HOPE) Score 1.meatus position 2.meatus shape 3.glans shape 4.penile skin shape 5.penile axis secreal 6.Torsion

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stock JA, Scherz HC, Kaplan GW. Distal hypospadias. Urol Clin North Am. 1995 Feb;22(1):131-8. PMID 7855949
- [Result] Elmoghazy H, Hussein MM, Mohamed E, Badawy A, Alsagheer G, Abd Elhamed AM. A novel technique for repair of mid-penile hypospadias using a preputial skin flap: results of 110 patients. Int Urol Nephrol. 2016 Dec;48(12):1943-1949. doi: 10.1007/s11255-016-1416-7. Epub 2016 Sep 13. PMID 27623810
- [Result] Nerli RB, Chandra S, Rai S, Dixit NS. Grafted tubularised incised plate: A right option in the management of failed mid-penile and distal hypospadias. Afr J Paediatr Surg. 2023 Jul-Sep;20(3):197-201. doi: 10.4103/ajps.ajps_19_22. PMID 37470555
- [Result] Holland AJ, Smith GH, Ross FI, Cass DT. HOSE: an objective scoring system for evaluating the results of hypospadias surgery. BJU Int. 2001 Aug;88(3):255-8. doi: 10.1046/j.1464-410x.2001.02280.x. PMID 11488741